CLINICAL TRIAL: NCT04265118
Title: Development of a Sideward Turning Beds to Treat Positional Obstructive Sleep Apnea
Brief Title: Sideward Turning Beds for Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SideBed
Record Dates: First submitted 2020-01-30; First posted 2020-02-11 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sideward Tilt of Bed (Experimental): During sleep, while lying in supine position, the participant will be tilted sidewards by the bed. In practice, the experimenter activates the bed at timepoints during the night where the participant is lying in supine position. Activating the bed results in one half of the bed lifting 10 to 40 Degrees sidewards.
  Interventions: Device: Sidewards Tilting Bed

INTERVENTIONS:
Device: Sidewards Tilting Bed — Sidewards tilting of the bed is hypothesized to induce a body position change in sleeping subjects.

SUMMARY:
The aim of this feasibility study is to compare different settings of a custom-made automated bed with respect to their ability to induce a change in the sleeping position of the user. In particular, it is of interest whether the bed mechanism is able to change the position of a user from supine to lateral position. At the same time, the investigators want to know whether the intervention provided by the bed results in an arousal in sleeping users. In addition, feasibility of detecting the position of the user using the un-obtrusive pressure sensors, which are integrated in the bed, will be assessed.

Within the experiment, the investigators will identify participants that are sleeping mainly in supine position by doing an acti-watch based screening measurement in their home setting. Those participants who are sleeping in supine position for more than 12.5% of the home recording with the acti-watch will be invited to come to the lab for one night measurement. The experimenter will trigger interventions of the bed manually when the participant is lying in supine position. The investigators will evaluate the position change using infrared cameras and the built in sensors of the bed. Furthermore, a commercially available home-measurement device to record polysomnography will be used to evaluate whether the intervention caused arousals.

DETAILED DESCRIPTION:
Obstructive positional sleep apnea

Obstructive sleep apnea (OSA) is characterised by a repetitive collapse of the upper airway during sleep, which results in apnea or hypopnoea associated with oxygen desaturations and arousals. OSA affects up to 30% of the adult male population, increases with age, and is associated with daytime sleepiness, increased risk of traffic accidents, arterial hypertension, vascular dysfunction and cardiovascular events. In 56% to 75% percent of these apnea patients, the apnea-hypopnea index is correlating with the body position. This subgroup of patients suffers from position-dependent sleep apnea, which is defined by a difference in the apnea hypopnea index between supine position and non-supine positions of at least 50%. Current treatment recommendation for OSA is continuous positive airway pressure (CPAP) ventilation, because of its potential beneficial impact on cardiovascular outcomes. However, a recent randomised controlled trial has not shown reduction in major cardiovascular endpoints in OSA patients with manifest cardiovascular disease allocated to CPAP. Therefore, the beneficial effect of CPAP treatment has been subject to extensive discussion recently. Furthermore, in mildly and moderately affected patients, compliance is sometimes limited due to various side effects. A valuable alternative, which has been suggested for these patients, is the so-called positional therapy. The aim of the therapy is to make the supine position uncomfortable so that patients actively avoid it. However, due to interruption of the sleep because of acoustic signals or an obstacle fixes at the patients back, current treatment options are associated with low long term compliance.

Mechanisms for turning a sleeping user sideward

In literature, several mechanisms have been proposed to shift the sleeping user of a bed form supine to lateral position. In general, these methods can be sorted into the following four categories:

1. Inclination of one side of the mattress
2. Tilting of the mattress around a middle axis
3. Using pressurized air chambers to reconfigure the mattress shape
4. Using vibration or disturbing stimuli as aversion therapy when the person is sleeping on the back Method number 4 does require active participation of the user and would therefore have the same limitations as conventional positional therapy. However, method 1 to 3 are promising candidates for an intelligent anti-sleep apnea bed.

Methods

In order to compare the three methods described above a custom-made automated bed that has a pressurized air-mattress and provides the ability either to incline half of the bed surface up to 70° or tilt the whole surface up to 45° was developed. The purpose of this study is to evaluate which of these three mechanisms is more effective in changing the position of the user from supine to lateral. Furthermore, the settings which are most likely to induce a position change will be determined. In addition, it will be evaluated which test settings cause the least arousals in sleeping users. Evaluating this in healthy participants is an important step on our way towards an intelligent bed for treatment of position dependent obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* 12.5 % of the sleep in the screening night spent in supine position.

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Injuries or pain that prevents sleeping in supine or lateral position.
* Pregnancy.
* Length longer than 2 m (larger than standard bed).
* investigators, their family members, employees and other dependent persons^.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-07-19 (Actual); Study Completion 2020-07-19 (Actual)

PRIMARY OUTCOMES:
Change in position of the upper body | 1 year
  Change in the position of the upper body in degree of turning around the longitudinal axis (derived from infrared Video and from bodyworn position sensor)
Arousals from sleep | 1 year
  Change of the orientation of the upper body assessed with the polysomnography device (asleep)

SECONDARY OUTCOMES:
Performance of the sensors | 1 year
  Accuracy, Sensitivity, Specificity of the pressure sensors in the matress

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riener, Prof. Dr., Principal Investigator — Swiss Federal Institute of Technology
Locations (1):
- SMS lab, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
We consider uploading the polysomnography data (electroencephalography, electromyography, electrooculography) of the night time measurements to the ETH Research Collection database to make them available to other investigators.
Supporting Information: CSR
Time Frame: The data will be ulpoaded to the research collection after study completion and is available there for a period of 15 years.
Access Criteria: Open Access
URL: https://www.research-collection.ethz.ch/